CLINICAL TRIAL: NCT06786338
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of SGB-9768 in Patients with Primary IgA Nephropathy, C3 Glomerulopathy, and Immune Complex-mediated Membranoproliferative Glomerulonephritis.
Brief Title: A Study of SGB-9768 in Patients with Complement-mediated Kidney Diseases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGB-9768-003
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: IgA Nephropathy (IgAN); C3 Glomerulopathy; IC-MPGN
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IgAN-1 (Experimental): 2 doses of SGB-9768 by subcutaneous (sc) injection
  Interventions: Drug: SGB-9768
- IgAN-2 (Experimental): 2 doses of SGB-9768 by subcutaneous (sc) injection
  Interventions: Drug: SGB-9768
- C3G/IC-MPGN (Experimental): 2 doses of SGB-9768 by subcutaneous (sc) injection
  Interventions: Drug: SGB-9768

INTERVENTIONS:
Drug: SGB-9768 — SGB-9768 for subcutaneous (SC) injection

SUMMARY:
This study looks at how well and safely SGB-9768 works for patients with certain kidney diseases: primary IgA nephropathy, C3 glomerulopathy, and immune complex-related membranoproliferative glomerulonephritis. It's a phase 2 trial done at several locations where both patients and doctors know what treatment is being given.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label study to evaluate of the efficacy and safety of SGB-9768 in patients with primary IgA nephropathy, C3 glomerulopathy, and immune complex-mediated membranoproliferative glomerulonephritis. The primary objective is to evaluate efficacy of SGB-9768 in reducing urine protein excretion and maintain kidney function in these patients. Secondly, safety, pharmacokinetics and pharmacodynamics will be charaterized.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Weight ≥40 kg, with a body mass index (BMI) between 15 and 35 kg/m²
* Biopsy-confirmed diagnosis of primary IgA nephropathy, C3 glomerulopathy or IC-MPGN, accompanied by C3 deposition in the glomeruli.
* Urine protein-to-creatinine ratio (UPCR) ≥0.75 g/g
* Estimated glomerular filtration rate (eGFR) (calculated using the CKD-EPI formula) must be ≥30 mL/min/1.73 m².
* Must be on a stable maximum tolerated doses of ACE inhibitors (ACEI) or angiotensin receptor blockers (ARB) for at least 12 weeks
* Participants of childbearing potential must use highly effective contraception during the study and for at least 12 weeks following the end of the study or last dose of study drug

Exclusion Criteria:

* Kidney biopsy indicates more than 50% tubular atrophy or interstitial fibrosis.
* Kidney biopsy shows more than 50% formation of glomerular crescents, or clinical signs suggestive of rapidly progressive glomerulonephritis.
* IgA nephropathy, C3 glomerulopathy, or IC-MPGN secondary to other diseases
* Presence of other systemic diseases or kidney diseases that may cause proteinuria
* Received immunosuppressants or other immunomodulators within 90 days prior to the first administration of the investigational drug
* Received B-cell targeted biologics or other biologics within 180 days prior to the first administration of the investigational drug
* Used SGLT2 inhibitors or endothelin receptor antagonists, unless have been stably used for 12 weeks or more
* Significant comorbidities
* History of any malignant tumors of any organ system within the past 5 years
* History of severe trauma or major surgery within 12 weeks prior to screening, or plans to undergo surgery during the study.
* History of immunodeficiency diseases, congenital asplenia or splenectomy.
* History of recurrent invasive infections, active systemic bacterial, viral, or fungal infections
* Positive test results for HBV, HCV, HIV
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 2.5 times the upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline in urine protein-creatinine ratio (UPCR) | 24 weeks

SECONDARY OUTCOMES:
change from baseline in UACR and 24h-urine protein | 24 weeks
change from baseline in estimated glomerular filtration rate (eGFR) | 36 weeks
Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs) | from erollment through week 36
Pharmacokinetics-Cmax | 24 hours
  Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics-Tmax | 24 hours
  Time at which the maximum plasma concentration (Cmax) occurs
Pharmacokinetics-AUClast | 24 hours
  Area under the plasma concentration-time curve from dosing (time zero) to the time of the last measured concentration
Pharmacokinetics-t1/2 | 24 hours
  Terminal Elimination Half-Life (t1/2)
Pharmacodynamics-C3 | baseline through week 36
  Change From Baseline in serum Complement 3 (C3) level
Pharmacodynamics-complement classical pathway activity by Wieslab® CP | baseline through week 36
  Change From Baseline in serum Complement Classical Pathway Activity
Pharmacodynamics-complement alternative pathway activity by Wieslab® AP | baseline through week 36
  Change From Baseline in Serum Complement Alternative Pathway Activity

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Guizhou Provincial People's Hospital, Guiyang
  - The affiliated hospital of Guizhou medical university, Guiyang
  - The first affiliated hospital, Zhejiang university school of medicine, Hangzhou
  - Huashan hospital, Shanghai
  - Northern Jiangsu People's Hospital, Yangzhou
  - General hospital of ningxia medical university, Yinchuan
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No